CLINICAL TRIAL: NCT02369705
Title: Diagnosis of Sleep-related Respiratory Disorders in Patients With Cardiac Disorders Such as Atrial Fibrillation, Heart Failure and Other Comorbidities
Brief Title: Validation of Ambulatory Sleep Test (WP200/U) Compared In-lab Sleep Testing in Cardiac Subjects
Status: Completed | Type: Observational
Sponsor: Itamar-Medical, Israel (Industry)
Responsible Party: Sponsor
Other Study IDs: WP200/U-Cardio-001
Record Dates: First submitted 2015-02-08; First posted 2015-02-24 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-04

CONDITIONS: Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Subjects with cardiac disorders will be tested in the sleep laboratory with a conventional full-night PSG recording along with WP 200/WP200U ambulatory sleep diagnostic device in a synchronized manner.

The PSG data will be scored manually by a trained polysomnographic scorer, according to standard criteria for this clinical routine.

The data obtained by the WP200/WP200U will be analyzed automatically for RDI, AHI, sleep stages, snoring (optional) and body position (optional), in addition to parameters specific to cardiac subjects. The analysis will be performed by the WP200/WP200U software (zzzPAT) and will be compared to the PSG's manual scoring which serves as a "Gold Standard".

DETAILED DESCRIPTION:
Subjects with cardiac disorders, referred to the sleep lab will be offered to participate in the study. Subjects will be asked to sign an informed consent form and will be screened for inclusion exclusion criteria.

Subject demographic and medical information will be acquired from the subject himself and/or from the subject's medical chart and will be recorded on the appropriate pre-study electronic case report forms.

The subjects will be admitted to the clinical sleep laboratory for one night, during which they will undergo conventional full night PSG recording with the standard PSG channels. The WP 200/WP200U wrist device, which includes the PAT and pulse oximeter probes will be worn on the wrist.

The investigator will not have access to the WP200/WP200U data while scoring the PSG data. During the study recording, the WP200/WP200U data will be recorded inside the device, without being displayed on the PSG monitor. Furthermore, the WP200/WP200U analysis is done automatically without knowledge of the PSG scoring results.

ELIGIBILITY:
Inclusion Criteria:

* Age between17-90
* Subject is able to read understand and sign the informed consent form.
* Subject with diagnosed cardiac disorders and/or other comorbidity
* Willing to sleep with the WP200/WP200U and PSG simultaneously in the sleep lab

Exclusion Criteria:

* Permanent pacemaker: atrial pacing or VVI without sinus rhythm
* Finger deformity that precludes adequate sensor appliance.
* Use of one of the following medications: alpha blockers, short acting nitrates (less than 3 hours before the study)

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with cardiac disorder, referred to the sleep lab for a night study, who consent to undergo an overnight sleep study in the clinical sleep laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of the WP200 and WP200U in assessing RDI, AHI, sleep stages compared to the "gold standard" - PSG | Within 1 year after data collection is complete.
  calculation of the sensitivity, specificity, agreement and correlation obtained by the WP200/WP200U device automatic-computerized analysis as compared to the manual scoring of the PSG that is considered the "gold standard" disorders for subjects with cardiac disorders and/or comorbidities, to the manual scoring of the PSG that serves as a "gold standard".

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Penzel, Prof., Principal Investigator — Charite University, Berlin, Germany; Richard Berry, Prof., Principal Investigator — University of Florida
Locations (10):
- United States (5):
  - Kaiser Los Angeles, Los Angeles, California
  - Kaiser Permanente Fontana, Los Angeles, California
  - Kaiser Permanente San Jose, San Jose, California
  - University of Florida, Gainsville, Florida
  - Stony Brook medical center sleep lab, Smithtown, New York
- Centre for sleep and Chronobiology, Toronto, Ontario, Canada
- Charité-Universitätsmedizin, Berlin, Germany
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Health Care Campus, Haifa
  - Ichilov Medical Center, Tel Aviv